CLINICAL TRIAL: NCT07352423
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Assess Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of ALXN2230 in Healthy Adult Participants
Brief Title: Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study of ALXN2230 in Healthy Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: R0689C00001; ALXN2230-HV-101 (Registry Identifier: Alexion)
Record Dates: First submitted 2026-01-12; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Healthy Adult Participants
Keywords: ALXN2230; Healthy Participants; Pharmacodynamics; Pharmacokinetics; PK; PD; Immunogenicity; First in Human; Single Ascending Dose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will be enrolled across multiple cohorts and will receive a single dose of placebo.
  Interventions: Drug: Placebo
- ALXN2230 (Experimental): Participants will be enrolled across multiple cohorts and will receive a single dose of ALXN2230.
  Interventions: Drug: ALXN2230

INTERVENTIONS:
Drug: ALXN2230 — Participants will receive ALXN2230 via SC injection. Optional cohort will receive ALXN2230 via SC infusion.
  Arms: ALXN2230
Drug: Placebo — Participants will receive placebo via SC injection. Optional cohort will receive placebo via SC infusion.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of single subcutaneous (SC) doses of ALXN2230 in healthy participants.

DETAILED DESCRIPTION:
Part A of this study is expected to enroll approximately 40 participants (30 on ALXN2230 and 10 on placebo) across 5 cohorts and Part B is expected to enroll approximately 8 participants (6 on ALXN2230 and 2 on placebo) in 1 cohort.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Baseline immunoglobulin G (IgG) concentrations ≥ 1000 milligrams per deciliter (mg/dL) and ≤ 1600 mg/dL at Screening.
* Antibody titers for Tetanus toxoid (≥ 0.1 International Units per milliliter (IU/mL)) at Screening.
* Nonsmokers and not using any nicotine-containing products. A nonsmoker is defined as an individual who has abstained from smoking for at least 1 year prior to Screening.
* BMI within the range 18 to 32 kilograms per square meter (kg/m2), inclusive; with body weight ≥ 50 kilograms (kg).

Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data.
* Abnormal blood pressure (BP) (resting BP not to exceed 140/80 mmHg and no less than 90/60 mmHg).
* Participants who have history of allergy or hypersensitivity to excipients in ALXN2230.
* History of unexplained, recurrent infection, or infection requiring treatment with systemic antibiotics within 90 days prior to dosing on Day 1.
* Pregnant or breastfeeding females are excluded from the clinical study.
* Participants with known clinically relevant immunological disorders.
* Lymphoma, leukemia, breast cancer or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 5 years.
* ALT > 1.0 × upper limit of normal (ULN)
* TBIL > 1.0 × ULN
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with exception for Gilbert's syndrome).
* QTc > 450 millisecond (msec) for male participants or > 470 msec for female participants.
* Significant blood loss (including blood donation [> 500 mL]) or had a transfusion of any blood product within 12 weeks prior to dosing or plan 1 within 4 weeks after the end of the study.

Additional inclusion/exclusion criteria may apply, per protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-02-24 (Estimated); Primary Completion 2026-12-23 (Estimated); Study Completion 2026-12-23 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs) | Day 1 up to Day 113

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of ALXN2230 | Day 1 up to Day 113
Time to Cmax (Tmax) of ALXN2230 | Day 1 up to Day 113
Area Under the Concentration-time Curve from Time 0 to the Last Quantifiable Concentration (AUCt) of ALXN2230 | Day 1 up to Day 113
Serum Concentration of Biomarkers | Day 1 up to Day 113

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a CSR synopsis and plain language summaries.
Supporting Information: CSR